CLINICAL TRIAL: NCT00396435
Title: Multicenter, Prospective, Randomised, Open-label Study, Evaluating the Effect of Two Levels of Haemoglobin on Quality of Life and Speed of Progression of Renal Insufficiency on Renal Transplanted Patients With Chronic Graft Dysfunction (CGD)
Brief Title: Correction of Anaemia and Progression of Renal Failure on Transplanted Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Centre Hospital-Universitaire d'Amiens, CHU
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPRIT
Record Dates: First submitted 2006-11-03; First posted 2006-11-07 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Anaemia; Renal Transplantation; Kidney Failure
Keywords: anaemia; renal transplantation; kidney failure
MeSH Terms: conditions — Anemia; Renal Insufficiency | interventions — epoetin beta; Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): High Hb target
  Interventions: Drug: Neorecormon
- Group B (Active Comparator): Low Hb Target
  Interventions: Drug: Neorecormon

INTERVENTIONS:
Drug: Neorecormon — Administration SC one a week in patients randomized in group A Administration SC if Hb below 10.5 g/dl in group B
  Other Names: Epoetin

SUMMARY:
The purpose of this study is to evaluate, on renal transplanted patients with CGD, the effect of two levels of haemoglobin on quality of life at 6 months and the speed of progression of renal function degradation at 24 months.

This study will recruit 140 patients in 21 centers in France.

DETAILED DESCRIPTION:
The number of patients arriving each year at the stage of final renal insufficiency (IRT) and requiring the dialysis of substitution does not cease growing, in parallel with continuous ageing of the population in industrialized countries. The incidence of the IRT is approximately 110 new patients per million inhabitants per year, which represents an annual progression from approximately 4% to 8% according to areas.Approximately 35000 patients are currently treated by dialysis, 90% by hemodialysis and 10% per peritoneal dialysis . The other alternative to the treatment of the IRT is renal transplantation. Approximately 2000 patients are transplanted each year in France, and it is estimated that a minimum of 3000 transplantations should annually be carried out in order to answer at the request of the patients registers on a chronic program of dialysis and in to be transplanted age.

The total number of patients living with a functional graft is approximately 15000.

The IRT is a major problem of public health and its cost is considerable: for less than 50000 patients, this one represents nearly 4% of the annual budget of the social security. To slow down the progression of the IRC represents a major therapeutic challenge, including at the transplanted patients.

The physiopathological mechanisms proposed to explain the harmful role of anaemia in the progression of the renal lesions during the IRC rest on the tissue hypoxia induced by the reduction in haemoglobin. The tissue hypoxia supports the development of the interstitial fibrosis by stimulating the production of type I collagen and some inhibitors of metalloproteases, implied in the extracellular matrix degradation. The hypoxia also stimulates the synthesis of TGF-beta, pro-fibrosing factors implied in the progression of many renal diseases, in particular the nephropathy diabetic. By reducing the hypoxia thanks to the correction of anaemia by the EPO, one can hope to slow down the progression of the interstitial fibrosis, and thus the progression of the renal insufficiency. Lastly, the correction of anaemia reduces resistance to insulin and the secondary hyperinsulinism to uraemia, improves the dyslipidemia and the oxidizing stress, factors also implied in the progression of many nephropathies, diabetic or not.

It appears that anaemia is a factor of risk of progression of the chronic nephropathies. To slow down the progression of the chronic dysfunction of the graft is an important challenge because of shortage of graft and impossibility, in the current state of the French centers of renal transplantation to carry out the number of necessary grafts to provide for the current waiting list. Our hypothesis, if it is checked, should make it possible to very appreciably improve the quality of life of the transplanted patients and to slow down the progression of their IRC, thus delaying the duration before return in dialysis.

Population: Renal patients transplanted since at least 12 months, presenting a CGD defined by 20 ml/mn/1,73 m2 > Clcr < 50 ml/mn/1,73 m2 and an anaemia (Hb < 11,5 g/dl)

The patients answering the criteria of selection will be assigned by randomization with the one of the two following groups:

* Group a: target haemoglobin: 13 to 15 g/dl
* Group b: target haemoglobin: 10,5 to 11,5 g/dl

Criteria of inclusion

* Adults of male or female sex of more than 18 years
* Patients having profited from one 1st or one the 2nd renal Transplantation
* Patients Transplanted since more than 1 year
* Patients having a CGD defined by Clcr < 50 ml/mn/1,73 m2
* Patients presenting an anaemia: Hb lower than 11,5 g/dl
* Absence of deficiency out of iron
* Patients having given their in writing consent

Study Treatment: Neorecormon® (Epoétine beta) under cutaneous injection

The objective of the study is to show a difference between group A "haemoglobin target: 13 to 15 g/dl" and group it B "haemoglobin target: 10,5 to 11,5 g/dl", with regard to the renal function.

The calculation of the number of patients is thus based on a model of covariance analysis in repeated measurements of clearance of creatinin on the whole of the times evaluated between J0 and M24 and on the following hypothesis:

* H0: no effect groups during the two years of follow-up
* H1: Effect groups, evolution different from the values of Clcr during the follow-up

The alfa-risk (probability of rejecting H0 wrongly) was fixed at 5% The beta-risk (probability of keeping H0 wrongly) at 10% The total number of patients to be randomized was estimated at 140 (70 by group) This number of patients will also make it possible to test the scores of quality of life with a power higher than 90%

ELIGIBILITY:
Inclusion Criteria:

* Adults male or female of 18 years male or female sex to 70 years
* Patients having profited from one 1st or one the 2nd transplantation
* Patients transplanted since more than 1 year and less than 20 years.
* Patients having a CDG defined by a clearance of creatinin, lower than 50 ml/mn/1,73 m2 (according to Gault and Cockcroft) and whose renal function is stable over the last 3 months (variation of Scr of less than 20% over the last 3 months)
* Patients presenting an anaemia: Hb lower than 11.5 g/dl
* No deficiency out of iron: Saturation of the transferrin > 20% and ironnemia > 50 mg/l at the time of the screening visit
* Patients having given their written consent

Exclusion Criteria:

* Major forms of drepanocytosis or thalassaemia
* Iron Deficit (CST < 20% or ferritin < 50 mg/l)
* Haemolysis (haptoglobin < 0,30 g/l)
* Severe renal insufficiency: Clcr < 20 ml/min/1,73 m2
* Severe Hyperparathyroidy (serum PTH > 800 pg/ml)
* Evolutionary chronic inflammatory Disease (CRP > 15 mg/l)
* Acute or chronic infectious disease
* Evolutionary neoplasic Disease
* Infection by the HIV and viral cirrhosis
* Recent Antecedents of MI or AIT (< 3 months)
* Severe Arteritis of the lower limbs (Stage III or IV)
* Acute Rejection requiring a treatment in the 3 previous months
* Blood Transfusion on the last 3 months
* Evolutionary GI Ulcer on the last 3 months
* Severe Arterial HyperTension not controlled by medicamentous treatment (NOT > 170 mm Hg or PAD > 100 mm Hg under treatment)
* Epilepsy of recent diagnosis
* Relevant biological value(at screening visit) : - Proteinuria > 3 g/24h
* Serum Albumin < 30 g/l
* Platelets > 600.000/µl
* Programmed heavy surgery
* Pregnancy or breast feeding
* Administration of an experimental drug in the 30 days preceding the screening visit
* Known Over-sensitiveness to Epoetin beta
* Patients under Sirolimus
* Patients under EPO at screening visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2004-04; Primary Completion 2009-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
eClcr by Cockcroft formula | 2 years

SECONDARY OUTCOMES:
Measure CDG by the clearance of Iohexol | 2 years
1/Scr at J0, 6 months, 12 months, 18 months and 24 months Scr with J0, 6, 12, 18 and 24 months | 2 years
Proteinuria and micro-albuminuria at J0, 12 and 24 months | 2 years
Evaluation of the quality of life in the 2 groups of patients per self-evaluation at J0 and 6 months | 6 months
Adverse events, in particular cardiovascular events: MI, AIT, Arteritis of lower limb, revascularisation, | 2 years
Biological tolerance: Albuminemia, pre-albuminemia, CRP, plasmatic Cholesterol, HDL and LDL | 2 years
Level of blood pressure at the beginning and the end of the study and comparison of the number of antihypertensive drugs received by patients before and after the 24 months of follow-up | 2 years
Number of units of beta-EPO managed in the 2 groups | 2 years
Number of patients receiving blood transfusions | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Choukroun, MD, PhD, Principal Investigator — CHU Amiens; Franck Martinez, MD, PhD, Principal Investigator — Hôpital Necker- Enfants Malades - PARIS
Locations (20):
- France (20):
  - Hôpital Sud, Amiens
  - Hôpital de Bois Guillaume, Bois-Guillaume
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Clémenceau, Caen
  - CHU Clermont Ferrand - Hôpital Gabriel Monpied, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - Hôpital de la Tronche, Grenoble
  - Hôpital Calmette, Lille
  - Hôpital Dupuytren, Limoges
  - Hôpital de la Conception, Marseille
  - Hôpital Pasteur, Nice
  - Hôpital Necker - Enfants Malades, Paris
  - Hôpital de la Milétrie, Poitiers
  - Hôpital Maison Blanche, Reims
  - Hôpital Pontchaillou, Rennes
  - Hôpital Civil, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpital Rangueil, Toulouse
  - CHU de Tours - Hôpital Bretonneau, Tours
  - Hôpital Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Choukroun G, Kamar N, Dussol B, Etienne I, Cassuto-Viguier E, Toupance O, Glowacki F, Moulin B, Lebranchu Y, Touchard G, Jaureguy M, Pallet N, Le Meur Y, Rostaing L, Martinez F; CAPRIT study Investigators. Correction of postkidney transplant anemia reduces progression of allograft nephropathy. J Am Soc Nephrol. 2012 Feb;23(2):360-8. doi: 10.1681/ASN.2011060546. Epub 2011 Dec 22. PMID 22193388
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280